CLINICAL TRIAL: NCT01111604
Title: An Open-label, Multicenter, Randomized Phase 2 Study Evaluating the Safety and Efficacy of 5 FU/FA and Oxaliplatin (Modified FOLFOX 6) in Combination With Ramucirumab or IMC-18F1 or Without Investigational Therapy as Second Line Therapy in Patients With Metastatic Colorectal Cancer Following Disease Progression on First Line Irinotecan-based Therapy
Brief Title: A Study of Ramucirumab or Icrucumab in Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13942; CP20-0801 (Other: ImClone Systems); I4Y-IE-JCDB (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-04-08; First posted 2010-04-27 (Estimated); Results first posted 2019-08-06 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2019-07

CONDITIONS: Colon Cancer; Rectal Cancer
Keywords: Colonic Neoplasms; Rectal Neoplasms; Adenocarcinoma; Antibodies, Monoclonal
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms; Adenocarcinoma | interventions — Ramucirumab; Icrucumab; IMC-18F1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- mFOLFOX-6 (Active Comparator): mFOLFOX-6
  Interventions: Drug: mFOLFOX-6
- mFOLFOX-6 + Ramucirumab (Experimental): mFOLFOX-6 + Ramucirumab
  Interventions: Biological: Ramucirumab; Drug: mFOLFOX-6
- mFOLFOX-6 + Icrucumab (Experimental): mFOLFOX-6 + Icrucumab
  Interventions: Biological: Icrucumab; Drug: mFOLFOX-6

INTERVENTIONS:
Biological: Ramucirumab — 8 mg/kg IV Q2W
  Other Names: IMC-1121B; LY3009806
  Arms: mFOLFOX-6 + Ramucirumab
Biological: Icrucumab — 15 mg/kg IV Q2W
  Other Names: IMC-18F1; LY3012212
  Arms: mFOLFOX-6 + Icrucumab
Drug: mFOLFOX-6 — Oxaliplatin: 85 milligram per square meter (mg/m²) IV every 2 weeks (Q2W)
  FA: 400 mg/m² IV Q2W (or LFA: 200 mg/m² Q2W if FA is unavailable).
  5FU: 400 mg/m² bolus + 2400 mg/m² IV Q2W

SUMMARY:
The purpose of this study is to determine if participants with metastatic colorectal cancer live longer without their cancer progressing when treated with standard chemotherapy, standard chemotherapy plus ramucirumab, or standard chemotherapy plus icrucumab.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the progression-free survival (PFS) in participants with metastatic colorectal cancer when treated with 1 of 3 modified FOLFOX-6 (folinic acid [FA] + fluorouracil [5-FU] + oxaliplatin [mFOLFOX-6])-based regimens, as second-line therapy.

During 2010, there has been an identified shortage of injectable folinic acid (FA) in the United States. Levo-folinic acid (LFA) will be allowed as a substitute for FA in the mFOLFOX-6 chemotherapy regimen in circumstances in which FA is not available, to facilitate continuity of participant care.

ELIGIBILITY:
Inclusion Criteria:

* Disease progression on an irinotecan-based first-line chemotherapy regimen (ie FOLFIRI or CAPIRI [capecitabine + irinotecan], with or without bevacizumab)
* Age ≥ 18 years
* Life expectancy of ≥ 6 months
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) 0-1 at study entry
* Agrees to adequate contraception during the study period and for 12 weeks after the last dose of study medication
* Provided signed informed consent

Exclusion Criteria:

* Has received prior oxaliplatin-based chemotherapy for locally advanced unresectable or metastatic Colorectal Cancer (CRC) (Prior oxaliplatin-based adjuvant chemotherapy is allowed if the last dose of oxaliplatin was administered > 12 months prior to randomization)
* Has documented and/or symptomatic brain or leptomeningeal metastases
* Has an ongoing or active infection, symptomatic or poorly controlled cardiac arrhythmia, psychiatric illness/social situations, or any other serious uncontrolled medical disorders
* On chronic non-topical corticosteroid treatment. A participant discontinuing such treatment > 3 months prior to randomization is eligible
* Has uncontrolled or poorly controlled hypertension on a standard regimen of antihypertensive therapy
* Has a concurrent active malignancy. A participant with previous history of malignancy is eligible, provided that he/she has been disease free for > 3 years
* If female, is pregnant (confirmed by serum beta human chorionic gonadotropin [βHCG] test) or lactating
* Has received a prior autologous or allogeneic organ or tissue transplantation
* Has undergone major surgery within 28 days prior to randomization
* Has had a serious nonhealing wound, ulcer, or bone fracture within 28 days prior to randomization
* Has an elective or planned major surgery to be performed during the course of the trial
* Has a history of inflammatory bowel disease requiring pharmacological and/or surgical intervention in the 12 months prior to randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2010-08; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (17):
- United States (3):
  - ImClone Investigational Site, Cincinnati, Ohio
  - ImClone Investigational Site, Columbia, South Carolina
  - ImClone Investigational Site, Nashville, Tennessee
- Canada (14):
  - ImClone Investigational Site, Calgary, Alberta
  - ImClone Investigational Site, Edmonton, Alberta
  - ImClone Investigational Site, Kelowna, British Columbia
  - ImClone Investigational Site, Surrey, British Columbia
  - ImClone Investigational Site, Vancouver, British Columbia
  - ImClone Investigational Site, Halifax, Nova Scotia
  - ImClone Investigational Site, Hamilton, Ontario
  - ImClone Investigational Site, London, Ontario
  - ImClone Investigational Site, Mississauga, Ontario
  - ImClone Investigational Site, Oshawa, Ontario
  - ImClone Investigational Site, Ottawa, Ontario
  - ImClone Investigational Site, Toronto, Ontario
  - ImClone Investigational Site, Windsor, Ontario
  - ImClone Investigational Site, Montreal, Quebec

REFERENCES:
- [Derived] Moore M, Gill S, Asmis T, Berry S, Burkes R, Zbuk K, Alcindor T, Jeyakumar A, Chan T, Rao S, Spratlin J, Tang PA, Rothenstein J, Chan E, Bendell J, Kudrik F, Kauh J, Tang S, Gao L, Kambhampati SR, Nasroulah F, Yang L, Ramdas N, Binder P, Strevel E. Randomized phase II study of modified FOLFOX-6 in combination with ramucirumab or icrucumab as second-line therapy in patients with metastatic colorectal cancer after disease progression on first-line irinotecan-based therapy. Ann Oncol. 2016 Dec;27(12):2216-2224. doi: 10.1093/annonc/mdw412. Epub 2016 Oct 11. PMID 27733377

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Completers were defined as participants who had failure event (progressive disease, death), or were off treatment and censored due to study completion.
Groups:
- mFOLFOX-6: mFOLFOX-6: Oxaliplatin: 85 milligram/meter squared, intravenous (mg/m², IV) infusion every 2 weeks (Q2W)
  Folinic acid (FA): 400 mg/m² IV infusion Q2W (or Levo-folinic acid [LFA]: 200 mg/m² Q2 weeks if FA is unavailable).
  Fluorouracil (5FU): 400 mg/m² bolus + 2400 mg/m² IV infusion Q2W
- mFOLFOX-6 + Ramucirumab: mFOLFOX-6 + Ramucirumab
  Ramucirumab: 8 mg/kg IV Q2W
  mFOLFOX-6: Oxaliplatin: 85 mg/m² IV Q2W
  FA: 400 mg/m² IV Q2W (or LFA: 200 mg/m² Q2W if FA is unavailable).
  5FU: 400 mg/m² bolus + 2400 mg/m² IV Q2W FA: 400 mg/m² IV infusion Q2 weeks (or LFA: 200 mg/m² Q2 weeks if FA is unavailable).
  5FU: 400 mg/m² bolus + 2400 mg/m² IV infusion Q2W
- mFOLFOX-6 + Icrucumab: mFOLFOX-6 + Icrucumab
  Icrucumab: 15 mg/kg IV Q2W
  mFOLFOX-6: Oxaliplatin: 85 mg/m² IV Q2W
  FA: 400 mg/m² IV Q2W (or LFA: 200 mg/m2 Q2W if FA is unavailable).
  5FU: 400 mg/m² bolus + 2400 mg/m² IV Q2W
  5FU: 400 mg/m² bolus + 2400 mg/m² IV Q2W
Period: Overall Study
Arm/Group | mFOLFOX-6 | mFOLFOX-6 + Ramucirumab | mFOLFOX-6 + Icrucumab
Started | 54 | 52 | 52
Received at Least One Dose of Study Drug | 49 | 52 | 52
Completed | 46 | 52 | 49
Not Completed | 8 | 0 | 3
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Withdrew Consent | 3 | 0 | 2
Not completed — Withdrawal by Subject | 2 | 0 | 0
Not completed — Death | 1 | 0 | 0
Not completed — Met Exclusion Criteria | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least one dose of study drug.
Groups:
- mFOLFOX-6: mFOLFOX-6: Oxaliplatin: 85 mg/m² IV Q2W
  FA: 400 mg/m² IV Q2W (or LFA: 200 mg/m² Q2W if FA is unavailable).
  5FU: 400 mg/m² bolus + 2400 mg/m² IV Q2W
- mFOLFOX-6 + Ramucirumab: mFOLFOX-6 + Ramucirumab
  Ramucirumab: 8 mg/kg IV Q2W
  mFOLFOX-6: Oxaliplatin: 85 mg/m² IV Q2W
  FA: 400 mg/m² IV Q2W (or LFA: 200 mg/m² Q2W if FA is unavailable).
  5FU: 400 mg/m² bolus + 2400 mg/m² IV Q2W
- mFOLFOX-6 + Icrucumab: mFOLFOX-6 + Icrucumab
  Icrucumab: 15 mg/kg IV Q2W
  mFOLFOX-6: Oxaliplatin: 85 mg/m² IV Q2W
  FA: 400 mg/m² IV Q2W (or LFA: 200 mg/m2 Q2W if FA is unavailable).
  5FU: 400 mg/m² bolus + 2400 mg/m² IV Q2W
- Total: Total of all reporting groups
Arm/Group | mFOLFOX-6 | mFOLFOX-6 + Ramucirumab | mFOLFOX-6 + Icrucumab | Total
Number analyzed (Participants) | 49 | 52 | 52 | 153
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.8 (9.23) | 59.9 (10.95) | 58.2 (10.15) | 59.6 (10.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 21 | 29 | 71
  Male | 28 | 31 | 23 | 82
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 49 | 52 | 51 | 152
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 7 | 5 | 7 | 19
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 3 | 1 | 0 | 4
  White | 35 | 45 | 45 | 125
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 3 | 0 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: PFS is defined as the time from baseline until the date of disease progression as defined by Response Evaluation Criteria in Solid Tumors (RECIST v1.1), or death from any cause, whichever was first. Participants who die without a reported prior progression will be considered to have progressed on the day of their death. Participants who did not progress, are lost to follow-up, or have missed two or more scheduled tumor assessments will be censored at the day of their last radiographic tumor assessment, if there are no post-baseline tumor measurements for a randomized and treated participant, the participant will be censored at the date of randomization. If death or progressive disease (PD) occurs after 2 or more missing radiographic visits, censoring will occur at the date of the last radiographic visit prior to the last visit.
Time Frame: Baseline until Disease Progression or Death from Any Cause (Up to 95 Weeks)
Population: Modified Intent-to-Treatment (mITT) population includes all the randomized participants who received at least one dose study drug. In mFOLFOX-6, mFOLFOX-6+Ramucirumab and mFOLFOX-6 + Icrucumab, there were 13, 9 and 11 censored participants, respectively.
Measure: Median (95% Confidence Interval); unit: Weeks
Groups:
- mFOLFOX-6: mFOLFOX-6: Oxaliplatin: 85 per meter squared (mg/m²) IV Q2W
  FA: 400 mg/m² IV Q2W (or LFA: 200 mg/m² Q2W if FA is unavailable).
  5FU: 400 mg/m² bolus + 2400 mg/m² IV Q2W
- mFOLFOX-6 + Ramucirumab: mFOLFOX-6 + Ramucirumab
  Ramucirumab: 8 mg/kg IV infusion Q2W
  mFOLFOX-6: Oxaliplatin: 85 mg/m² IV Q2W
  FA: 400 mg/m² IV Q2W (or LFA: 200 mg/m² Q2W if FA is unavailable).
  5FU: 400 mg/m² bolus + 2400 mg/m² IV Q2W
- mFOLFOX-6 + Icrucumab: mFOLFOX-6 + Icrucumab
  Icrucumab: 15 mg/kg IV Q2W
  mFOLFOX-6: Oxaliplatin: 85 mg/m² IV infusion Q2W
  FA: 400 mg/m² IV infusion Q2 weeks (or LFA: 200 mg/m² Q2W if FA is unavailable).
  5FU: 400 mg/m² bolus + 2400 mg/m² IV Q2W
Arm/Group | mFOLFOX-6 | mFOLFOX-6 + Ramucirumab | mFOLFOX-6 + Icrucumab
Number analyzed (Participants) | 49 | 52 | 52
Weeks | 18.4 [15.7 to 24.4] | 21.4 [16.1 to 25.0] | 15.9 [14.1 to 16.4]

2. Secondary Outcome: Percentage of Participants Achieving Complete Response (CR) or Partial Response (PR) (Objective Response Rate [ORR])
Description: The ORR is the percentage of participants with Complete Response (CR, the disappearance of target lesions and any pathological lymph nodes [target or non-target] taking as reference the baseline sum of diameters in response to treatment) or Partial Response (PR, at least a 30% decrease in the sum of diameter of target lesions, taking as reference the baseline sum diameters in response to treatment) according to RECIST v1.1 from the start of the treatment until disease progression.
Time Frame: Baseline until Disease Progression (Up to 95 Weeks)
Population: mITT population includes all the randomized participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- mFOLFOX-6: mFOLFOX-6
  mFOLFOX-6: Oxaliplatin: 85 mg/m² IV Q2W
  FA: 400 mg/m² IV Q2W (or LFA: 200 mg/m² Q2W if FA is unavailable).
  5FU: 400 mg/m² bolus + 2400 mg/m² IV Q2W
- mFOLFOX-6 + Ramucirumab: mFOLFOX-6 + Ramucirumab
  Ramucirumab: 8 mg/kg IV Q2W
  mFOLFOX-6: Oxaliplatin: 85 mg/m² IV Q2W
  FA: 400 mg/m² I.V. infusion q2 weeks (or LFA: 200 mg/m² Q2W if FA is unavailable).
  5FU: 400 mg/m² bolus + 2400 mg/m² IV Q2W
- mFOLFOX-6 + Icrucumab: mFOLFOX-6 + Icrucumab
  Icrucumab: 15 mg/kg IV Q2W
  mFOLFOX-6: Oxaliplatin: 85 mg/m² IV Q2W
  FA: 400 mg/m² I.V. infusion q2 weeks (or LFA: 200 mg/m² Q2W if FA is unavailable).
  5FU: 400 mg/m² bolus + 2400 mg/m² I.V. infusion Q2W
Arm/Group | mFOLFOX-6 | mFOLFOX-6 + Ramucirumab | mFOLFOX-6 + Icrucumab
Number analyzed (Participants) | 49 | 52 | 52
percentage of participants | 14 [5.94 to 27.24] | 3.8 [0.47 to 13.21] | 3.8 [0.47 to 13.21]

3. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is defined as the time from baseline to the date of death from any cause. If the participant is alive at the end of the follow-up period or is lost to follow-up, OS will be censored on the last date the participant is known to be alive.
Time Frame: Baseline Until Death from Any Cause (Up to 163 Weeks)
Population: mITT population includes all the randomized participants who received at least one dose of study drug. In mFOLFOX-6, mFOLFOX-6 + Ramucirumab, and mFOLFOX-6 + Icrucumab there were 12, 11, and 12 censored participants, respectively.
Measure: Median (95% Confidence Interval); unit: Weeks
Groups:
- mFOLFOX-6: mFOLFOX-6
  mFOLFOX-6: Oxaliplatin: 85 per meter squared (mg/m²) IV Q2W
  FA: 400 mg/m² IV Q2W (or LFA: 200 mg/m² Q2W if FA is unavailable).
  5FU: 400 mg/m² bolus + 2400 mg/m² IV Q2W
- mFOLFOX-6 + Icrucumab: mFOLFOX-6 + Icrucumab
  Icrucumab: 15 mg/kg IV Q2W
  mFOLFOX-6: Oxaliplatin: 85 mg/m² IV Q2W
  FA: 400 mg/m² IV Q2W (or LFA: 200 mg/m² Q2W if FA is unavailable).
  5FU: 400 mg/m² bolus + 2400 mg/m² IV Q2W
Arm/Group | mFOLFOX-6 | mFOLFOX-6 + Ramucirumab | mFOLFOX-6 + Icrucumab
Number analyzed (Participants) | 49 | 52 | 52
Weeks | 53.6 [36.1 to 68.4] | 41.7 [28.4 to 60.3] | 42.0 [32.0 to 50.4]

4. Secondary Outcome: Duration of Response (DoR)
Description: DoR was measured from the time measurement criteria are first met for Complete Response or Partial Response or until the first date that the criteria for disease progression or death from any cause. whichever is first recorded. As defined according to RECIST v1.1, CR is the disappearance of all non-nodal target lesions, and PR is the short axes of any target lymph nodes reduced to < 10 mm and at least a 30% decrease in the sum of the diameters of target lesions including the short axes of any target lymph nodes.)
Time Frame: Criteria First Met for CR or PR until Disease Progression or Death from Any Cause (Up to 95 Weeks)
Population: mITT population includes all the randomized participants who received at least one dose of study drug and had evaluable baseline and post baseline DoR data. 2 participants were censored in mFOLFOX-6 arm, 2 in mFOLFOX-6 + Ramucirumab arm and 1 in mFOLFOX-6 + Icrucumab.
Measure: Median (95% Confidence Interval); unit: Weeks
Groups:
- mFOLFOX-6: mFOLFOX-6: Oxaliplatin: 85 mg/m² IV Q2W
  FA: 400 mg/m² IV Q2W(or LFA: 200 mg/m² Q2W if FA is unavailable).
  5FU: 400 mg/m² bolus + 2400 mg/m² IV infusion Q2W
- mFOLFOX-6 + Ramucirumab: mFOLFOX-6 + Ramucirumab
  IMC-1121B: 8 mg/kg IV Q2W
  mFOLFOX-6: Oxaliplatin: 85 mg/m² IV Q2W
  FA: 400 mg/m² IV Q2W (or LFA: 200 mg/m² Q2W if FA is unavailable).
  5FU: 400 mg/m² bolus + 2400 mg/m² IV Q2W
- mFOLFOX-6 + Icrucumab: mFOLFOX-6 + Icrucumab
  IMC-18F1: 15 mg/kg IV Q2W
  mFOLFOX-6: Oxaliplatin: 85 mg/m² IV Q2W
  FA: 400 mg/m² IV Q2W (or LFA: 200 mg/m² Q2W if FA is unavailable).
  5FU: 400 mg/m² bolus + 2400 mg/m² IV Q2W
Arm/Group | mFOLFOX-6 | mFOLFOX-6 + Ramucirumab | mFOLFOX-6 + Icrucumab
Number analyzed (Participants) | 7 | 2 | 2
Weeks | 35.6 [4.0 to NA] — NA= data not evaluable by Kaplan-Meier method due to sample size of participants | NA [NA to NA] — N of 2 participants were censored therefore no evaluable data was collected. | NA [8.1 to NA] — N of 1 participant was censored therefore only individual data is presented, 8.1 weeks.

5. Secondary Outcome: Pharmacokinetics (PK): Maximum Concentration (Cmax) at Cycle 5
Description: Maximum concentration (1 hour post end of infusion, Cmax) is the concentration measured in serum.
Time Frame: Cycle 5, 1 Hour Post End of Infusion
Population: All randomized participants assigned to the mFOLFOX-6 + Ramucirumab or mFOLFOX-6 + Icrucumab who received at least one dose of study drug and had evaluable ramucirumab or icrucumab PK data to calculate Cmax.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram/milliliter (µg/mL)
Groups:
- mFOLFOX-6 + Ramucirumab: mFOLFOX-6 + Ramucirumab
  IMC-1121B: 8 mg/kg IV Q2W mFOLFOX-6: Oxaliplatin: 85 mg/m² IV Q2W
  FA: 400 mg/m² I.V. infusion q2 weeks (or LFA: 200 mg/m² Q2W if FA is unavailable).
  5FU: 400 mg/m² bolus + 2400 mg/m² IV Q2W
- mFOLFOX-6 + Icrucumab: mFOLFOX-6 + Icrucumab
  IMC-18F1: 15 mg/kg IV Q2W
  mFOLFOX-6: Oxaliplatin: 85 mg/m² IV Q2W
  FA: 400 mg/m² I.V. infusion q2 weeks (or LFA: 200 mg/m² Q2W if FA is unavailable).
  5FU: 400 mg/m² bolus + 2400 mg/m² IV Q2W
Arm/Group | mFOLFOX-6 + Ramucirumab | mFOLFOX-6 + Icrucumab
Number analyzed (Participants) | 2 | 3
microgram/milliliter (µg/mL) | NA (NA) — Geometric mean and Coefficient of Variation were not calculated because number of participants was <3. Values equal 12.900/54.5000 (min/max) | 201 (88)

6. Secondary Outcome: Pharmacokinetics (PK): Trough Serum Concentrations (Ctrough) at Cycle 5
Description: Trough (prior to infusion, Ctrough) concentrations measured in serum.
Time Frame: Cycle 5, Prior to Infusion
Population: All randomized participants assigned to the mFOLFOX-6 + Ramucirumab or mFOLFOX-6 + Icrucumab who received at least one dose of study drug and had evaluable Ramucirumab or Icrucumab PK data to calculate Ctrough.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | mFOLFOX-6 + Ramucirumab | mFOLFOX-6 + Icrucumab
Number analyzed (Participants) | 3 | 4
µg/mL | 53.6 (123) | 146 (32)

7. Secondary Outcome: Maximum Concentration (Cmax) at Day 8
Description: Maximum concentration (Cmax) is the maximum peak concentration measured in blood plasma after drug infusion.
Time Frame: Day 8 (cycles 1 and 5)
Population: Zero participants analyzed. Outcome Measure (OM) entered incorrectly and no data collected to report.
Arm/Group | mFOLFOX-6 + Ramucirumab | mFOLFOX-6 + Icrucumab
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Maximum Concentration (Cmax) at Day 15
Description: Cmax is the maximum peak concentration measured in blood plasma after drug infusion.
Time Frame: Day 15 (Cycles 1 and 5)
Population: Zero participants analyzed. OM entered incorrectly and no data collected to report.
Arm/Group | mFOLFOX-6 + Ramucirumab | mFOLFOX-6 + Icrucumab
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Minimum Concentration (Cmin) at Day 1
Description: Cmin is the minimum peak concentration measured in blood plasma after drug infusion.
Time Frame: Day 1 (cycles 1, 5, 9, and 13)
Population: Zero participants analyzed. OM entered incorrectly and no data collected to report.
Arm/Group | mFOLFOX-6 + Ramucirumab | mFOLFOX-6 + Icrucumab
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Minimum Concentration (Cmin) at Day 4
Description: Cmin is the minimum peak concentration measured in blood plasma after drug infusion.
Time Frame: Day 4 (cycles 1 and 5)
Population: Zero participants analyzed. OM entered incorrectly and no data collected to report.
Arm/Group | mFOLFOX-6 + Ramucirumab | mFOLFOX-6 + Icrucumab
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Minimum Concentration (Cmin) at Day 8
Description: Minimum concentration (Cmin) is the minimum peak concentration measured in blood plasma after drug infusion.
Time Frame: Day 8 (cycles 1 and 5)
Population: Zero participants analyzed. OM entered incorrectly and no data collected to report.
Arm/Group | mFOLFOX-6 + Ramucirumab | mFOLFOX-6 + Icrucumab
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Minimum Concentration (Cmin) at Day 15
Description: Minimum concentration (Cmin) is the minimum peak concentration measured in blood plasma after drug infusion.
Time Frame: Day 15 (cycles 1 and 5)
Population: Zero participants analyzed. OM entered incorrectly and no data collected to report.
Arm/Group | mFOLFOX-6 + Ramucirumab | mFOLFOX-6 + Icrucumab
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Number of Participants With Serum Ramucirumab Antibody Assessment
Description: A sample will be considered positive for anti-Ramucirumab antibodies if it exhibits a post-baseline antibody level exceeding the normal anti-Ramucirumab antibody level seen in healthy untreated individuals.
Time Frame: 31 Weeks
Population: Participants in mFOLFOX-6 +Ramucirumab who received at least one dose of study drug and had at least 1 post treatment assessment.
Measure: Count of Participants; unit: Participants
Groups:
- mFOLFOX-6 + Ramucirumab: mFOLFOX-6 + Ramucirumab
  Ramucirumab: 8 mg/kg IV Q2W
  mFOLFOX-6: Oxaliplatin: 85 mg/m² IV Q2W
  FA: 400 mg/m² I.V. infusion q2 weeks (or LFA: 200 mg/m² Q2W if FA is unavailable).
  5FU: 400 mg/m² bolus + 2400 mg/m² I.V. infusion q2 weeks
Arm/Group | mFOLFOX-6 + Ramucirumab
Number analyzed (Participants) | 52
Participants | 0

14. Secondary Outcome: Serum Anti-Icrucumab Antibody Assessment
Description: A sample will be considered positive for anti-icrucumab antibodies if it exhibits a post-baseline antibody level exceeding the normal anti-icrucumab antibody level seen in healthy untreated individuals.
Time Frame: 31 Weeks
Population: Zero participants analyzed. No data collected to report.
Groups:
- mFOLFOX-6 + Icrucumab: mFOLFOX-6 + Icrucumab
  Icrucumab: 15 mg/kg IV Q2W
  mFOLFOX-6: Oxaliplatin: 85 mg/m² IV Q2W
  FA: 400 mg/m² IV Q2W (or LFA: 200 mg/m² Q2W if FA is unavailable).
  5FU: 400 mg/m² bolus + 2400 mg/m² I.V. infusion Q2W
Arm/Group | mFOLFOX-6 + Icrucumab
Number analyzed (Participants) | 0

15. Secondary Outcome: Number of Participants With Adverse Events
Description: A summary of serious AEs (SAEs) and all other non-serious AEs regardless of causality, is located in the Reported Adverse Events module.
Time Frame: Baseline up to 165 weeks
Population: Population includes all the randomized participants who received at least one dose study drug.
Measure: Count of Participants; unit: Participants
Groups:
- mFOLFOX-6: mFOLFOX-6
  mFOLFOX-6: Oxaliplatin: 85 mg/m² I.V. infusion q2 weeks
  FA: 400 mg/m² I.V. infusion q2 weeks (or LFA: 200 mg/m2 q2 weeks if FA is unavailable).
  5FU: 400 mg/m² bolus + 2400 mg/m² I.V. infusion q2 weeks
- mFOLFOX-6 + Ramucirumab: mFOLFOX-6 + Ramucirumab
  IMC-1121B: 8 mg/kg I.V. infusion, administered every 2 weeks
  mFOLFOX-6: Oxaliplatin: 85 mg/m² I.V. infusion q2 weeks
  FA: 400 mg/m² I.V. infusion q2 weeks (or LFA: 200 mg/m2 q2 weeks if FA is unavailable).
  5FU: 400 mg/m² bolus + 2400 mg/m² I.V. infusion q2 weeks
- mFOLFOX-6 + Icrucumab: mFOLFOX-6 + Icrucumab Icrucumab: 15 mg/kg I.V. infusion, administered every 2 weeks mFOLFOX-6: Oxaliplatin: 85 mg/m² I.V. infusion q2 weeks FA: 400 mg/m² I.V. infusion q2 weeks (or LFA: 200 mg/m2 q2 weeks if FA is unavailable).
  5FU: 400 mg/m² bolus + 2400 mg/m² I.V. infusion q2 weeks
Arm/Group | mFOLFOX-6 | mFOLFOX-6 + Ramucirumab | mFOLFOX-6 + Icrucumab
Number analyzed (Participants) | 49 | 52 | 52
Participants
  Any TEAE | 49 | 52 | 52
  Any SAE | 11 | 18 | 12
  Any Grade ≥3 AE | 30 | 37 | 31
  Any AE leading to discontinuation (any drug) | 6 | 18 | 11

ADVERSE EVENTS:
Description: All randomized participants who received at least one dose of study drug.
Groups:
- mFOLFOX-6 + Ramucirumab: mFOLFOX-6 + Ramucirumab
  Ramucirumab : 8 mg/kg I.V. infusion, administered every 2 weeks
  mFOLFOX-6: Oxaliplatin: 85 mg/m² I.V. infusion q2 weeks
  FA: 400 mg/m² I.V. infusion q2 weeks (or LFA: 200 mg/m2 q2 weeks if FA is unavailable).
  5FU: 400 mg/m² bolus + 2400 mg/m² I.V. infusion q2 weeks
Arm/Group | mFOLFOX-6 | mFOLFOX-6 + Ramucirumab | mFOLFOX-6 + Icrucumab
All-Cause Mortality (participants affected / at risk) | 37/49 | 41/52 | 40/52
Serious Adverse Events (participants affected / at risk) | 11/49 | 18/52 | 12/52
Other Adverse Events (participants affected / at risk) | 48/49 | 52/52 | 52/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | mFOLFOX-6 (N=49) | mFOLFOX-6 + Ramucirumab (N=52) | mFOLFOX-6 + Icrucumab (N=52)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Peritonitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2)
Fatigue (General disorders) | 0 (0) | 2 (2) | 1 (1)
Infusion related reaction (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 3 (3)
Bile duct obstruction (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0)
Bile duct stenosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Neutropenic infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Medication error (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Stent occlusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Nephrotic syndrome (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Ureteric obstruction (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Embolism (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | mFOLFOX-6 (N=49) | mFOLFOX-6 + Ramucirumab (N=52) | mFOLFOX-6 + Icrucumab (N=52)
Anaemia (Blood and lymphatic system disorders) | 9 (12) | 7 (19) | 12 (33)
Neutropenia (Blood and lymphatic system disorders) | 16 (37) | 16 (39) | 12 (19)
Thrombocytopenia (Blood and lymphatic system disorders) | 12 (35) | 9 (37) | 3 (5)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 3 (4)
Lacrimation increased (Eye disorders) | 3 (4) | 2 (2) | 8 (9)
Vision blurred (Eye disorders) | 2 (2) | 1 (1) | 5 (6)
Abdominal distension (Gastrointestinal disorders) | 3 (3) | 6 (10) | 9 (10)
Abdominal pain (Gastrointestinal disorders) | 13 (21) | 16 (20) | 24 (37)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0)
Ascites (Gastrointestinal disorders) | 2 (2) | 6 (11) | 8 (9)
Constipation (Gastrointestinal disorders) | 12 (21) | 18 (27) | 19 (32)
Diarrhoea (Gastrointestinal disorders) | 19 (53) | 30 (54) | 27 (68)
Dry mouth (Gastrointestinal disorders) | 2 (5) | 3 (3) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 7 (11) | 2 (2) | 1 (1)
Flatulence (Gastrointestinal disorders) | 2 (2) | 0 (0) | 6 (6)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 4 (4) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 5 (5) | 2 (3)
Nausea (Gastrointestinal disorders) | 30 (61) | 24 (42) | 36 (82)
Proctalgia (Gastrointestinal disorders) | 5 (5) | 2 (2) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 12 (30) | 19 (30) | 12 (19)
Toothache (Gastrointestinal disorders) | 0 (0) | 6 (6) | 1 (1)
Vomiting (Gastrointestinal disorders) | 17 (31) | 13 (21) | 27 (58)
Asthenia (General disorders) | 0 (0) | 5 (6) | 2 (2)
Chills (General disorders) | 4 (4) | 1 (1) | 2 (2)
Face oedema (General disorders) | 0 (0) | 2 (2) | 13 (15)
Fatigue (General disorders) | 35 (86) | 45 (91) | 36 (106)
Infusion related reaction (General disorders) | 5 (19) | 7 (9) | 3 (7)
Mucosal inflammation (General disorders) | 1 (1) | 3 (3) | 0 (0)
Non-cardiac chest pain (General disorders) | 2 (2) | 3 (5) | 1 (1)
Oedema peripheral (General disorders) | 5 (13) | 15 (28) | 29 (54)
Pyrexia (General disorders) | 11 (12) | 9 (13) | 8 (11)
Temperature intolerance (General disorders) | 21 (76) | 13 (33) | 18 (66)
Oral candidiasis (Infections and infestations) | 0 (0) | 3 (4) | 2 (2)
Sinusitis (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 5 (5) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 3 (4) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 6 (7) | 3 (6) | 4 (8)
Blood alkaline phosphatase increased (Investigations) | 6 (10) | 5 (7) | 2 (5)
Lymphocyte count decreased (Investigations) | 2 (9) | 1 (3) | 3 (14)
Neutrophil count decreased (Investigations) | 7 (12) | 5 (9) | 5 (7)
Platelet count decreased (Investigations) | 3 (16) | 8 (50) | 4 (10)
Weight decreased (Investigations) | 7 (8) | 14 (18) | 4 (9)
White blood cell count decreased (Investigations) | 3 (8) | 4 (6) | 3 (6)
Anorexia (Metabolism and nutrition disorders) | 16 (29) | 20 (26) | 27 (46)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 1 (2) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 3 (4) | 6 (13) | 6 (9)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (4) | 3 (3) | 2 (4)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 (7) | 4 (7) | 7 (16)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (5) | 3 (3) | 9 (14)
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 (8) | 2 (2) | 6 (6)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (5) | 4 (10) | 3 (7)
Hypophosphataemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 2 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 3 (4) | 6 (10)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (14) | 8 (9) | 7 (11)
Flank pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (3) | 3 (5)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (3) | 4 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (7) | 1 (2) | 1 (1)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 5 (9) | 0 (0) | 3 (8)
Dizziness (Nervous system disorders) | 2 (3) | 7 (9) | 6 (6)
Dysaesthesia (Nervous system disorders) | 3 (5) | 7 (27) | 4 (6)
Dysgeusia (Nervous system disorders) | 5 (5) | 6 (9) | 17 (21)
Headache (Nervous system disorders) | 8 (12) | 16 (29) | 9 (12)
Memory impairment (Nervous system disorders) | 1 (2) | 3 (3) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 12 (22) | 12 (23) | 10 (13)
Paraesthesia (Nervous system disorders) | 2 (4) | 3 (11) | 5 (6)
Peripheral sensory neuropathy (Nervous system disorders) | 27 (94) | 25 (72) | 32 (81)
Depression (Psychiatric disorders) | 0 (0) | 3 (3) | 1 (1)
Insomnia (Psychiatric disorders) | 7 (8) | 7 (8) | 10 (13)
Proteinuria (Renal and urinary disorders) | 1 (1) | 6 (11) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (10) | 16 (19) | 10 (11)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 4 (7) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 10 (13) | 16 (20)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 2 (2) | 3 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 14 (17) | 3 (5)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 3 (4)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 6 (6)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2) | 2 (3)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 3 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (6) | 0 (0) | 1 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (4) | 1 (1) | 5 (5)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 4 (10)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 3 (5) | 6 (10) | 1 (1)
Periorbital oedema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 6 (7)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (4) | 4 (5) | 2 (3)
Rash (Skin and subcutaneous tissue disorders) | 3 (5) | 15 (22) | 8 (9)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 3 (4) | 3 (3) | 1 (2)
Flushing (Vascular disorders) | 1 (1) | 2 (3) | 3 (3)
Hypertension (Vascular disorders) | 1 (1) | 15 (24) | 5 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days